CLINICAL TRIAL: NCT01871116
Title: A Randomized Study Evaluating the Effect of a Remote-Based Weight Loss Program (POWER-remote) on Biomarkers in Women With Early Stage Breast Cancer
Brief Title: POWER-remote Weight Loss Program in Early Stage Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J12128; J12128 (Other: SKCCC at Johns Hopkins)
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Early Stage Breast Cancer
Keywords: breast cancer; early stage; weight loss
MeSH Terms: conditions — Breast Neoplasms; Weight Loss

STUDY DESIGN:
Intervention Model Description: Weight loss intervention versus self-directed weight loss.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- POWER-remote (Experimental): Participants will start a weight loss program called POWER-remote for Breast Cancer Survivors. This program involves two main components: an online portion accessed on a computer through the internet and a telephone portion to help monitor progress.
  Interventions: Behavioral: POWER-remote
- Self-directed (Active Comparator): Participants will receive a pamphlet entitled "Aim for a Healthy Weight", to help guide weight loss goals without access to the web-based POWER-remote system and coach support.
  Interventions: Behavioral: Self-directed

INTERVENTIONS:
Behavioral: POWER-remote — Web-based weight loss program.
  Arms: POWER-remote
Behavioral: Self-directed — Pamphlet entitled "Aim for a Healthy Weight" will be given.
  Arms: Self-directed

SUMMARY:
This research is being done to assess the effectiveness of a weight loss program in women with early stage breast cancer whose body mass index (BMI) is in the overweight or obese range (>25). Weight loss is beneficial in improving cardiovascular risk factors and overall health, but may also decrease the chance of breast cancer coming back. A weight loss counseling program was studied in a general population and was found to be effective to help reduce weight over a 2 year period.

The main goal of this study is to determine if women with a recent diagnosis of early breast cancer will also lose weight with this program. To better understand the effect that weight loss has on women with breast cancer, we will compare the patterns in blood and breast tissue samples (tissue biopsies will be optional), and questionnaires evaluating different aspects of one's well-being, before and after a dietary intervention or no intervention.

DETAILED DESCRIPTION:
The prevalence of obesity has increased rapidly in recent years. Epidemiological studies since the 1970's have strongly suggested that excess body weight gain may be a major risk factor for many cancers including breast cancer. In addition, once diagnosed with breast cancer, women who are overweight or obese experience worse outcomes despite standard local and adjuvant therapy. Furthermore, most women gain weight following a diagnosis of breast cancer, and this weight gain may increase risk of recurrence by 40-50% and breast cancer-related mortality by 53-60%.

A great deal of effort has been made for many years to explain the relationship between obesity and breast cancer. Molecularly, the relationship involves dynamic and complex interactions between a milieu of hormones, cytokines, adipokines, affecting cell signaling and potentially epigenetic pathways. Recently, studies in postmenopausal women have shown that weight loss modulates these cytokines and adipokines favorably. Inflammation associated with obesity can also be characterized pathologically when macrophages surround necrotic adipocytes in what are called crown-like structures (CLS). Furthermore, increased central obesity as measured by waist-to-hip ratios, may be associated with hypermethylation of certain breast cancer genes, and physical activity can reduce methylation of certain breast cancer-associated genes.

The Women's Intervention Nutrition Study (WINS) demonstrated that women with early-stage breast cancer receiving conventional cancer management randomized to a dietary intervention group had lower risk of relapse compared to those in a control group in those who lost weight. While women with a diagnosis of breast cancer are therefore recommended to maintain ideal body weight, limited progress has been made in developing feasible weight loss programs. However, collaborators from the Welch Center for Prevention, Epidemiology, and Clinical Research at the Johns Hopkins University have recently reported impressive and sustained weight loss in randomized controlled trials designated Practice-based Opportunities for Weight Reduction (POWER) in obese women with at least one cardiovascular risk factor using a remote-support weight loss intervention.

The overall goal of this study is to determine the effectiveness of the remote-support weight loss intervention of the POWER study, designated POWER-remote, in women with early breast cancer who are overweight or obese, and to assess the effects of weight loss of ≥5% body weight at 6 months and on biomarkers associated with obesity, inflammation, and breast cancer. The data will be used to implement a clinical intervention available to all overweight and obese women with breast cancer, and to design definitive studies assessing the impact of weight loss and biomarker modulation on risk of recurrent disease or development of new primary breast cancers.

ELIGIBILITY:
Inclusion Criteria:

* Women
* 18 years or older
* Ductal carcinoma in situ (DCIS) or stage I-III invasive breast cancer
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Current BMI ≥ 25 kg/m2 and weight ≤ 400 lbs, and willing to lose >5% of their body weight. NOTE: Participants may not have documented weight loss greater than 5% of body weight from time of diagnosis. Exceptions that are felt to be due to surgical or other procedures (e.g., mastectomies or reconstruction) may be allowed with prior approval of the Protocol Chair/designee.
* Patients must have completed local therapy (i.e. surgery and radiation therapy), and any preoperative or adjuvant chemotherapy within >3 and <60 months of registration. NOTE: Concurrent anti-HER2 therapy is permitted. Concurrent endocrine breast cancer therapy is permitted; patients may enroll >3 months after initiation of hormone therapy if expected to continue the same hormone agent for at least the first 6 months of the study. Concurrent enrollment in other interventional or drug clinical trials is at the discretion of the Protocol Chair.
* Willingness to change diet, physical activity and weight.
* To ensure compliance with the POWER-remote and PatientViewpoint programs, patients must meet the following: prior experience with web forms and feels able to use the POWER-remote web program and PatientViewpoint; has or is able to download Internet Explorer 8+, Firefox 3.0+, Safari 4.0+, Chrome 4.0+, and Adobe Flash Player 10; familiarity with and access to internet at least 4 days per week; use of an email program or willing and able to establish one for this study; and, able to read and write the English language without assistance.
* Patient is aware of her diagnosis, understands the study regimen, its requirements, risks, and discomforts, and is able and willing to sign an informed consent form.

Exclusion Criteria:

* History of another prior cancer within the last 5 years, with the exception of another breast cancer, adequately treated cone-biopsied in situ carcinoma of the cervix uteri, and basal or squamous cell carcinoma of the skin
* Medical condition likely to hinder accurate measurement of weight, including any condition: for which weight loss is contraindicated, which would likely cause weight loss, or which would affect adipokine and inflammatory markers (e.g., end stage renal disease (ESRD) on dialysis, cirrhosis, autoimmune disease, adrenal disease, and history of bariatric surgery).
* The use of the following medications are excluded: insulin or sulfonylureas; patients with thyroid disease who are not on stable doses of thyroid medication for at least the past 6 months; medications that cause weight loss (e.g., topiramate, bupropion, exenatide, lorcaserin, phentermine or orlistat) within the past 3 months; medications that are likely to cause weight gain or prevent weight loss (e.g., corticosteroids, lithium, olanzapine, risperidone, clozapine, oral contraceptive pills, hormone replacement therapy) within the past 3 months; medications that may affect adipokine or inflammatory markers (e.g., sulfonylureas, glitazones, insulin, steroids, ACE inhibitors, beta blockers and statins) unless started ≥3 months prior to enrollment, or chronic NSAIDS (defined as use of ≥3 times a week) for ≥1 month.
* Pregnant or nursing within past 6 months, or plans to become pregnant in the next year
* Currently enrolled or planning to enroll in a weight loss program (e.g., Innergy, Weight Watchers, Jenny Craig, Nutrisystem, and Medifast).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in body weight | After 12 months
  To compare the proportion of women with early stage breast cancer, who have completed all local therapy and adjuvant chemotherapy, who lose ≥5% of their baseline body weight after 6 and 12 months between a control arm (self-directed weight loss) and an experimental arm (POWER-remote)

SECONDARY OUTCOMES:
Change in biomarkers | After 12 months
  To evaluate the effects of weight loss and POWER-remote on serum biomarkers (including fasting glucose, fasting lipids, fasting insulin, insulin like growth factor (IGF), high-sensitivity C-reactive protein (hsCRP), interleukin 1 and 6 (IL-1 and IL-6), tumor necrosis factor- alpha (TNF-α), leptin, adiponectin, and estradiol) at baseline and 6 months
Change in PROs (Patient Reported Outcomes) | After 12 months
  To evaluate the effects of weight loss and POWER-remote on PROs, with a specific interest in comparing the change in Physical Function at 6 months from baseline as a function of weight los

CONTACTS AND LOCATIONS:
Overall Officials: Vered Stearns, M.D., Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
All participant data is deidentified and will be grouped together when presenting results.

REFERENCES:
- [Derived] Sheng JY, Chen R, Rosner GL, Snyder CF, Appel LJ, Stearns V, Smith MT, Coughlin JW. The Impact of Baseline Sleep as a Potential Moderator of Weight Loss Intervention in Breast Cancer Survivors: Results From the POWER-Remote Trial. Obesity (Silver Spring). 2025 Dec 15. doi: 10.1002/oby.70096. Online ahead of print. PMID 41397701